CLINICAL TRIAL: NCT01670084
Title: A Phase II Study of Combination Nilotinib and Hyper-CVAD in Patients Newly Diagnosed With Philadelphia-Chromosome Positive Acute Lymphoblastic Leukemia or Chronic Myeloid Leukemia Blast-Phase Lymphoid Lineage
Brief Title: Nilotinib and Combination Chemotherapy in Treating Patients With Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia or Blastic Phase Chronic Myelogenous Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1184; NCI-2012-01061 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Philadelphia Chromosome Positive Adult Precursor Acute Lymphoblastic Leukemia; Untreated Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Methotrexate; merphos; Cytarabine; Prednisone; Mesna; Dexamethasone; Calcium Dobesilate; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nilotinib, combination chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: nilotinib; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: methotrexate; Drug: cytarabine; Drug: prednisone; Drug: mesna; Drug: dexamethasone; Drug: leucovorin calcium

INTERVENTIONS:
Drug: nilotinib — Given PO
  Other Names: AMN 107; Tasigna
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: methotrexate — Given IV or IT
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: cytarabine — Given IV or IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Drug: mesna — Given IV
  Other Names: mercaptoethane sulfonate; Mesnex; MSA
Drug: dexamethasone — Given IV or PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV

SUMMARY:
In this study researchers want to find out more about the side effects of a new drug for Philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia (ALL) and chronic myelogenous leukemia (CML) blastic phase (BP) and if this disease will respond better to nilotinib combined with standard hyper-CVAD therapy rather than hyper-CVAD alone. Hyper-CVAD is a combination of cyclophosphamide, mesna, vincristine (vincristine sulfate), doxorubicin (doxorubicin hydrochloride), dexamethasone, methotrexate, cytarabine, and rituximab (only for patients with cluster of differentiation [CD]20 positive disease). Researchers don't know all the ways that this drug may affect people

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical efficacy (2-year disease-free survival rate) of nilotinib and combination chemotherapy in adult patients newly diagnosed with Philadelphia chromosome positive B-cell acute lymphoblastic leukemia or blast crisis of chronic myeloid leukemia.

SECONDARY OBJECTIVES:

I. Determine the 2-year overall survival rate. II. Determine the complete response (CR) rates (hematological, cytogenetic, and molecular) in patients treated with this regimen.

III. Determine the CR duration in patients treated with this regimen. IV. Assess the safety and toxicity of this regimen by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

TERTIARY OBJECTIVES:

I. Assess the prognostic and predictive factors for patients treated with this regimen.

II. Assess the cerebrospinal fluid (CSF) penetration for Nilotinib (CSF Nilotinib levels) in humans.

III. Assess the Abelson (ABL) kinase domain mutations frequency at diagnosis, during therapy, and at relapse.

OUTLINE:

INDUCTION AND CONSOLIDATION SCHEDULE A (COURSES 1, 3, 5, 7): Patients receive cyclophosphamide intravenously (IV) twice daily (BID) over 2 hours on days 1-3, mesna IV continuously on days 1-3, doxorubicin hydrochloride IV push on day 4, vincristine sulfate IV on days 4 and 11, dexamethasone IV or orally (PO) on days 1-4 and 11-14, methotrexate intrathecally (IT) on day 2, cytarabine IT on day 8, and nilotinib PO BID on days 1-14. Patients with CD20-positive disease also receive rituximab IV on days 1 and 11.

INDUCTION AND CONSOLIDATION SCHEDULE B (COURSES 2, 4, 6, 8): Patients receive methotrexate IV continuously over 24 hours on day 1, cytarabine IV over 2 hours on days 2-3, leucovorin calcium IV every 6 hours on days 2-3, methotrexate IT on day 2, cytarabine IT on day 8, and nilotinib PO BID on days 1-14. Patients with CD20-positive disease also receive rituximab IV on days 1 and 11.

MAINTENANCE (COURSES 9-32): Patients receive nilotinib PO BID on days 1-28 (days 1-14 for minimal residual disease [MRD]-positive patients), vincristine sulfate IV on day 1, and prednisone PO on days 1 to 5. Patients also receive rituximab IV on day 1 of each course if CD20-positive, every sixth course if MRD-negative, or every third course if MRD-positive.

INTENSIFICATION: Patients receive treatment as in Schedule A in courses 14 and 21 of maintenance therapy and treatment as in Schedule B in courses 15 and 22 of maintenance therapy.

DELAYED MAINTENANCE (COURSES 33-36): Patients receive nilotinib PO BID on days 1 to 84. Treatment repeats every 84 days for up to 4 courses.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, histological confirmed Philadelphia positive B-cell acute lymphoblastic leukemia or chronic myeloid leukemia blast-phase lymphoid lineage (bilineal, biphenotypic or undifferentiated) per World Health Organization (WHO) criteria; NOTE: Dexamethasone (or corticosteroids) use is allowed if needed before starting chemotherapy; prior imatinib or dasatinib therapy for CML chronic phase (CP) or accelerated phase (AP) is allowed
* Molecular or cytogenetic documentation of BCR-ABL fusion gene via any of the following: reverse transcriptase-polymerase chain reaction (RT-PCR), G-banding, or fluorescence in situ hybridization (FISH) testing from peripheral blood and/or bone marrow sampling
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Magnesium/potassium/phosphorus within normal limits (WNL)
* Serum amylase =< 1.5 x upper limit of normal (ULN)
* Lipase =< 1.5 x ULN
* Total bilirubin < 1.5 x ULN (does not apply to patients with isolated hyperbilirubinemia [e.g., Gilbert's disease], in this situation the direct bilirubin =< 2 x ULN)
* Alkaline phosphatase =< 3 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN
* Creatinine =< 1.5 x ULN
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to return to Mayo Clinic Rochester or Mayo Clinic Arizona for follow-up during the active monitoring phase of the study
* Willing to provide CSF and blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following because this study involves investigational agent(s) whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the study and for 3 months after completion of study treatment
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive (even if on highly active antiretroviral therapy [HAART])
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
* History of myocardial infarction =< 12 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Previous treatment with chemotherapy or any other tyrosine kinase inhibitor (prior imatinib or dasatinib for CML-CP/-AP is allowed)
* Impaired cardiac function including any one of the following:

  * Inability to monitor the QT interval on electrocardiogram (ECG)
  * Congenital long QT syndrome or a known family history of long QT syndrome
  * Cardiac ejection fraction (EF) < 45%
  * Clinically significant resting brachycardia (< 50 beats per minute)
  * Corrected QT interval (QTc) > 450 msec on baseline ECG; if QTc > 450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
  * Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension)
  * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
* Patients receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450 3A4 (CYP3A4); use of the following strong or moderate inhibitors are prohibited =< 7 days prior to registration:

  * Strong Inhibitors of CYP3A4; > 5-fold increase in the plasma area under the curve (AUC) values or more than 80% decrease in clearance

    * Indinavir (Crixivan®)
    * Nelfinavir (Viracept®)
    * Atazanavir (Reyataz®)
    * Ritonavir (Norvir®)
    * Clarithromycin (Biaxin®, Biaxin XL®)
    * Itraconazole (Sporanox®)
    * Ketoconazole (Nizoral®)
    * Nefazodone (Serzone®)
    * Saquinavir (Fortovase®, Invirase®)
    * Telithromycin (Ketek®)
  * Moderate Inhibitors of CYP3A4; > 2-fold increase in the plasma AUC values or 50-80% decrease in clearance

    * Aprepitant (Emend®)
    * Erythromycin (Erythrocin®, E.E.S. ®, Ery-Tab®, Eryc®, EryPed®, PCE®)
    * Fluconazole (Diflucan®)
    * Grapefruit juice
    * Verapamil (Calan®, Calan SR®, Covera-HS®, Isoptin SR®, Verelan®, Verelan PM®)
    * Diltiazem (Cardizem®, Cardizem CD®, Cardizem LA®, Cardizem SR®, Cartia XT™, Dilacor XR®, Diltia XT®, Taztia XT™, Tiazac®)
* Patients receiving any medications or substances that are inducers of CYP3A4; use of the following inducers are prohibited =< 7 days prior to registration

  * Inducers of CYP3A4
  * Efavirenz (Sustiva®)
  * Nevirapine (Viramune®)
  * Carbamazepine (Carbatrol®, Epitol®, Equetro™, Tegretol®, Tegretol-XR®)
  * Modafinil (Provigil®)
  * Phenobarbital (Luminal®)
  * Phenytoin (Dilantin®, Phenytek®)
  * Pioglitazone (Actos®)
  * Rifabutin (Mycobutin®)
  * Rifampin (Rifadin®)
  * St. John's wort
* Patients currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery)
* Acute or chronic pancreatic disease
* Known cytopathologically confirmed central nervous system (CNS) infiltration
* Acute or chronic liver disease or severe renal disease considered unrelated to the cancer
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Major surgery =< 4 weeks prior to registration or not recovered from prior surgery
* Treatment with other investigational agents =< 14 days of registration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate, defined as a patient who is alive and relapse-free, in patients who achieve a CR during the first 2 courses out to 2 years | 2 years
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Overall survival time, defined as the time from registration to death due to any cause out to 2 years | 2 years
Complete response (CR) rate estimated by the number of patients achieving an objective status of CR during the first 2 courses of treatment divided by the total number of evaluable patients | 56 days
Complete response (CR) as defined for all evaluable patients who have achieved a CR as the date at which the patient's objective status is first noted to be a CR to the earliest date relapse is documented out to 4 years | Up to 4 years
Maximum grade for each type of adverse event, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Up to 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Aref Al-Kali, M.D., Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota